CLINICAL TRIAL: NCT04868708
Title: A Multicenter, Open-label, Phase II Study of AK104（an Anti-PD-1 and Anti-CTLA-4 Bispecific Antibody) in the Treatment of Recurrent or Metastatic Cervical Cancer
Brief Title: A Study of AK104（ an Anti-PD-1 and Anti-CTLA-4 Bispecific Antibody) in Recurrent or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK104-210
Record Dates: First submitted 2021-04-05; First posted 2021-05-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Recurrent or Metastatic Cervical Cancer
Keywords: immuno-oncology; an Anti-PD-1 and Anti-CTLA-4 Bispecific Antibody; Recurrent or metastatic cervical cancer; PD-1; CTLA-4
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Bevacizumab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK104+Paclitaxel+Cisplatin/Carboplatin (Experimental): AK104 intravenously(IV) every 3 weeks (Q3W)
  Paclitaxel 175mg/m2 IV every 3 weeks (Q3W)
  Cisplatin 50mg/m2 or Carboplatin AUC5 IV every 3 weeks (Q3W)
  Interventions: Biological: AK104; Drug: Paclitaxel; Drug: Cisplatin or Carboplatin
- AK104+Bevacizumab+Paclitaxel+Cisplatin/Carboplatin (Experimental): AK104 every 3 weeks (Q3W)
  Bevacizumab 15mg/kg IV every 3 weeks (Q3W)
  Paclitaxel 175mg/m2 IV every 3 weeks (Q3W)
  Cisplatin 50mg/m2 or Carboplatin AUC5 IV every 3 weeks (Q3W)
  Interventions: Biological: AK104; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin or Carboplatin
- AK104 (Experimental): AK104 IV every 2 weeks (Q2W)
  Interventions: Biological: AK104

INTERVENTIONS:
Biological: AK104 — Subjects will receive AK104 intravenously.
Biological: Bevacizumab — Subjects will receive Bevacizumab intravenously.
  Arms: AK104+Bevacizumab+Paclitaxel+Cisplatin/Carboplatin
Drug: Paclitaxel — Subjects will receive Paclitaxel intravenously.
  Other Names: PTX
  Arms: AK104+Bevacizumab+Paclitaxel+Cisplatin/Carboplatin; AK104+Paclitaxel+Cisplatin/Carboplatin
Drug: Cisplatin or Carboplatin — Subjects will receive Cisplatin or Carboplatin intravenously.
  Other Names: DDP,CBP
  Arms: AK104+Bevacizumab+Paclitaxel+Cisplatin/Carboplatin; AK104+Paclitaxel+Cisplatin/Carboplatin

SUMMARY:
This is a multicenter, open-label, phase II clinical study conducted in China. All subjects will receive AK104 in combination with standard treatment regimens or AK104 alone. The primary end point is safety. The secondary end point is efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
* Estimated life expectancy of ≥3 months.
* Histologically or cytologically confirmed recurrent or metastatic cervical cancer that not appropriate for radical surgical resection and/or radical radiotherapy or chemotherapy.
* For cohort A and B: The pathological types were squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma. No previous systematic treatment for recurrent or metastatic cervical cancer.
* For cohort C: The pathological types were squamous cell carcinoma or adenosquamous cell carcinoma. Subjects must have received platinum-containing dual-drug chemotherapy combination with bevacizumab during or after the recurrence or metastasis phase and have demonstrated radiologically confirmed disease progression during or after treatment. Subjects will have no more than 2 lines of systemic therapy in the recurrence or metastatic stages.
* Subjects must have at least one measurable lesion in accordance with RECIST v1.1.
* All subjects must provide archived or freshly acquired tumor tissue samples, approximately 5 unstained FFPE pathological slides.
* Adequate organ function.
* Females of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first administration. If having sex with an unsterilized male partner, the subject must use an acceptable contraceptive method since screening and must agree to continue using this contraceptive method for 120 days after the last administration.

Exclusion Criteria:

* Subjects had clinically significant hydronephrosis that could not be relieved by nephrostomy or urethral stenting, as determined by the investigator.
* Other active malignancies within 2 years prior to the first administration. Subjects with locally curable tumors that appear to be cured, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the breast, were not excluded.
* Have received other study drugs or study devices within 4 weeks prior to the first administration.
* Is participating in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period for an interventional study.
* Subjects received systemic treatment with either proprietary Chinese drugs with anti-tumor indications or herbal medicines with anti-tumor effects, or immunomodulatory drugs (thymopeptide, interferon, interleukin) within 2 weeks prior to the first administration.
* Had received the last course of systemic antitumor therapy within 4 weeks prior to the first administration; Underwent major surgery within 3 weeks; Received non-specific immunoregulatory system treatment within 2 weeks; Any herbal or proprietary Chinese medicine with anti-tumor indications was received within 2 weeks.
* Have previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as antibodies targeting ICOS, CD40, CD137, GITR, and Ox40 targets, etc.), immune cell therapy, etc. Any treatment targeted at the immune mechanism of tumor.
* Subjects had an active autoimmune disease that required systemic treatment within 2 years prior to the first administration, or an autoimmune disease that was determined by the investigator to be likely to recur or for which treatment was planned.
* Active or documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis, or chronic diarrhea).Inability to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal disorders that can seriously affect the administration and absorption of drug.
* Subjects requiring systemic treatment with glucocorticoids (> 10 mg/ day equivalent dose of prednisone) or other immunosuppressive agents within 14 days prior to the first administration.
* Known history of Immunodeficiency.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Underwent major surgery or severe trauma within 28 days prior to the first administration; Underwent surgery to improve or reduce the risk of tumor complications within 14 days prior to the first administration; Or have not fully recovered from previous surgery. Significant surgery is planned within 30 days after the first administration (as determined by the investigator).
* Medical history of gastrointestinal perforation, gastrointestinal fistula, and female reproductive tract fistula within 6 months prior to the first administration; If the perforation or fistula has been treated by excision or repair and the disease has been recovered or remitted as determined by the investigator, admission is allowed.
* Known history of interstitial lung disease.
* Known history of active tuberculosis (TB).
* Serious infections within 4 weeks prior to the first administration, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
* An active infection requiring systemic therapy.
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 1000 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <1000 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Known history of testing positive for human immunodeficiency virus (HIV).
* Metastases of the central nervous system, metastases of pia mater, spinal cord compression, or pia mater disease confirmed by imaging or pathological examination.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Clinically active hemoptysis, active diverticulitis, peritoneal abscess, or gastrointestinal obstruction.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria.
* Grade ≥2 peripheral nerve disease, defined according to the NCI CTCAE V5.0 standard.
* Receipt of live or attenuated vaccination within 30 days prior to the first administration, or plan to receive live or attenuated vaccine during the study.
* Known history of serious hypersensitivity reaction to other monoclonal antibodies.
* Subjects with known contraindications to cisplatin/carboplatin, paclitaxel and bevacizumab or a history of allergy/hypersensitivity to any of their components (refer to the relevant drug label, not applicable for Cohort C, bevacizumab-related contraindications and allergy to bevacizumab only to Cohort B).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
AE | From the time of informed consent signed through 90 days after the last dose of AK104
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK104 until death due to any cause.
Minimum observed concentration (Cmin) of AK104 at steady state | From first dose of AK104 through 30 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK105 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 30 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Expression of PD-L1 in tumor tissue samples | Baseline (Tumor tissue samples must be provided to the research center or central laboratory prior to initial administration)
  PD-L1 expression will be determined by IHC in the central laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD, Principal Investigator — Hunan Cancer Hospital; Hanmei Lou, Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lou H, Cai H, Huang X, Li G, Wang L, Liu F, Qin W, Liu T, Liu W, Wang ZM, Li B, Xia Y, Wang J. Cadonilimab Combined with Chemotherapy with or without Bevacizumab as First-Line Treatment in Recurrent or Metastatic Cervical Cancer (COMPASSION-13): A Phase 2 Study. Clin Cancer Res. 2024 Apr 15;30(8):1501-1508. doi: 10.1158/1078-0432.CCR-23-3162. PMID 38372727
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38372727/